CLINICAL TRIAL: NCT06573437
Title: Clinical Performance of the VESTO® Vascular Stent for Treatment of Iliac Peripheral Obstructive Arterial Disease - Post Market Clinical Trial Iliac Stent Trial
Brief Title: Clinical Performance of the VESTO® Vascular Stent for Treatment of Iliac Peripheral Obstructive Arterial Disease
Acronym: VESTO-ILIAC
Status: Recruiting | Type: Observational
Sponsor: Braile Biomedica Ind. Com. e Repr. Ltda. (Industry)
Responsible Party: Sponsor
Other Study IDs: VESTO PMCF - Iliac Stent trial
Record Dates: First submitted 2024-08-21; First posted 2024-08-27 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2024-08

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Vascular Stent - Vesto Endoprosthesis — Vascular Stent Implant - Vesto Endoprosthesis

SUMMARY:
This study will validate the efficacy and safety of the VESTO® Vascular Stent for treating patients with iliac peripheral arterial obstructive disease in a post-market clinical trial

DETAILED DESCRIPTION:
Multicenter study aimed at collecting post-market clinical data on the VESTO® vascular stent for the treatment of patients with iliac peripheral arterial occlusive disease requiring endovascular intervention. The objective of the study is to evaluate the short-term (12-month) safety and clinical performance of the Vesto® vascular stent in patients with iliac peripheral arterial occlusive disease.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older;
2. TASC-II aortoiliac lesion classification of modified class A, B, C, or D;
3. Rutherford classification score of 2 to 5;
4. Access site compatibility with the device delivery system;
5. Compliance with the device's instructions for use (IFU);
6. Patient availability for appropriate follow-up times for the duration of the study;
7. Patient informed about the nature of the study, agreeing to its provisions, and signing the informed consent form.

Exclusion Criteria:

1. Known hypersensitivity to heparin, contrast media, or stent components;
2. Patient with blood dyscrasia;
3. Pregnant or breastfeeding women;
4. Patient currently participating in an investigational drug or device study;
5. Patient undergoing chemotherapy or radiation therapy;
6. Patient with a stent or graft located in the target limb;
7. Patient who underwent angioplasty or bypass surgery within 30 days prior to inclusion in this study;
8. Patient with a life expectancy of less than 12 months;
9. Inability to undergo dual antiplatelet therapy (DAPT)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with iliac peripheral artery obstructive disease requiring endovascular treatment.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-06-21 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of Device-Related Serious Adverse Events (Device Safety) | 30 days post-index procedure
  Absence of major serious adverse events occurring within 30 days after the index procedure, defined as device- or procedure-related death, acute myocardial infarction (AMI), or above-the-metatarsal amputation in the treated leg due to a vascular event
Number of Patients with Technical Success (Device Performance) | Intraoperative
  Technical success with the absence of serious adverse events related to the device
Number of Patients Without Rupture or Dissection of the Treated Vessel (Combined Safety and Performance Outcome) | 30 days post index procedure
  Absence of rupture or dissection of the treated vessel within 30 days after the procedure

SECONDARY OUTCOMES:
Rate of Technical Success | Intraoperative
  Defined as the successful deployment of the endoprosthesis at the intended site with patency and absence of significant device deformities (e.g., kinks, stent eversion, twisting)
Rate of Procedural Success | 30 days post index procedure
  Defined as the absence of serious adverse events related to the device within 30 days
Incidence of Adverse Events | 30 days, 3, 6, 9, and 12 months
  Defined as device- or procedure-related death, bleeding or hematoma, myocardial infarction (MI), thrombosis, arterial rupture or dissection, or amputation above the metatarsal in the treated leg due to a vascular event
Conversion Rate to Open Surgery | Intraoperative
  Rate of patients who required conversion to open surgery
Primary Patency Rate | 30 days post index procedure
  Defined as the absence of restenosis > 50% within 30 days
Number of Patients with Clinical Success | 30 days, 3, 6, 9, and 12 months
  Defined by symptom improvement
Rate of Target Vessel Patency | 3, 6, 9, and 12 months
  Absence of restenosis > 50%
Limb Salvage Rate | 30 days, 6, 9, and 12 months
  When patients with rest pain experienced pain relief and those with foot ulcers showed improved perfusion, avoiding the need for amputation
Need for Endovascular Reintervention at the Target Lesion | 30 days, 3, 6, 9, and 12 months
  Percentage of patients who required additional endovascular procedures at the same anatomical site as the initial intervention

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Cypreste Oliveira, Principal Investigator — Hospital Santa Helena
Locations (6):
- Brazil (6):
  - Hospital Ana Nery, Salvador, Estado de Bahia
  - Hospital Santa Helena, Goiânia, Goiás
  - Hospital Universitário Pedro Ernesto (HUPE-UERJ), Rio de Janeiro, Rio de Janeiro
  - HCFMB-UNESP - Hospital das Clínicas da Faculdade de Medicina de Botucatu da Universidade Estadual Paulista, Botucatu, São Paulo
  - Hospital de Clínicas da Universidade Estadual de Campinas, Campinas, São Paulo
  - Hospital das Clínicas da Faculdade de Medicina de Ribeirão Preto, Ribeirão Preto, São Paulo

IPD SHARING:
Plan to Share IPD: No